CLINICAL TRIAL: NCT03801941
Title: Cross Over Pilot Study for Evaluation of Pain Reduction in Patients With Chronic Low Back Pain (for More Than 3 Month) Using an Innovative Handheld Device
Brief Title: Alleviating Trunk Low Back Pain, With an Active Medical Device Study (ATLAS)
Acronym: ATLAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Japet Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2016_67; 2018-A01729-46 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2019-01-03; First posted 2019-01-14 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Chronic Low Back Pain
Keywords: Low back pain; Medical device; Spine; Rehabilitation; Traction
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Wearing the ATLAS device 60 min per day during 5 days and evaluation of pain during standardized activities with the ATLAS Device at the 4th day and without the device at the 5th day of a 4 weeks rehabilitation program.
  Interventions: Device: wearing ATLAS device during evaluation at 4th day; Other: wearing ATLAS device during evaluation at 5th day
- Group B (Experimental): Wearing the ATLAS device 60 min per day during 5 days and evaluation of pain during standardized activities without the ATLAS Device at the 4th day and with the device at the 5th day of a 4 weeks rehabilitation program.
  Interventions: Device: wearing ATLAS device during evaluation at 4th day; Other: wearing ATLAS device during evaluation at 5th day

INTERVENTIONS:
Device: wearing ATLAS device during evaluation at 4th day — Wearing the ATLAS device 60 min per day during 5 days and evaluation of pain during standardized activities with or without ATLAS Device at the 4th or 5th day of a 4 weeks rehabilitation program.
Other: wearing ATLAS device during evaluation at 5th day — Wearing the ATLAS device 60 min per day during 5 days and evaluation of pain during standardized activities without ATLAS Device at the 4th or 5th day of a 4 weeks rehabilitation program.

SUMMARY:
The aim of the study is to evaluate the reduction of pain by wearing the ATLAS Medical Device in standardized daily activities for patients with Chronic Low Back Pain.

This is an intervention al non blinded study with a crossover design comparing pain evaluated with an Analogue Visual Scale with and without the ATLAS device during 5 standardized daily activities.

DETAILED DESCRIPTION:
This study aims at assessing pain release by wearing a new medical device (ATLAS) in patients affected by chronic low back pain.

Population: patients with chronic low back pain admitted for a 4 weeks rehabilitation program.

Intervention: active rehabilitation and wearing the ATLAS device 60 min per day. The ATLAS study is carried out during the 5 first days of the rehabilitation program.

Primary outcome: Pain intensity evaluation with a 100 mm Visual Analogue Scale (VAS) during 5 standardized activities (the most intensive pain during the 5 activities is recorded), with and without wearing the ATLAS device.

Secondary outcome measures: percentage of patients reporting pain decrease of at least 20 mm on the 100 mm VAS during the 5 standardized activities with the ATLAs device compared without wearing the device. Percentage of relieved patients (percentage of patient reporting pain intensity less than 30 mm on the 100 mm VAS with wearing the device). Pain intensity evaluated with the 100 mm VAS before and after 60 min of wearing the ATLAS device.

Randomization: two groups (i.e. group A and B). Primary outcome is evaluated at day 4 and 5, with a crossover design (Group A: pain is evaluated during activities with the device at day 4 and without the device at day 5. Group B: pain is evaluated during activities without the device at day 4 and with the device at day 5).

ELIGIBILITY:
Inclusion Criteria:

* Chronic low back pain for more than 3 month
* Analogical visual scale superior or egal to 3/10
* BMI < 30
* 18 < Age < 75 years
* Patients who signed the informed consent
* Hospital Anxiety and depression score less than 11

Exclusion Criteria:

* - Neurological or radicular deficit
* Skin pathology of the trunk region
* Antecedent of surgery of spinal fusion
* Implanted neurostimulation treatment
* Scoliosis with Cobb angle > 30°
* History of vertebral fracture
* BMI > 30
* Respiratory failure
* Recent rib fracture (less than 3 month)
* Pregnancy or breastfeeding
* Osteoporosis
* Refusal to participate to the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Pain release with the ATLAS device during standardized daily activities | at 5th day of a 4 weeks rehabilitation program.
  Pain intensity evaluation with a 100 mm Visual Analogue Scale (VAS) from 0 to 100 mm (0 means no pain and 100 means extremely severe pain) during the standardized daily activities (the most intense pain reported during the 5 activities is recorded).

SECONDARY OUTCOMES:
Pain release with the ATLAS device during standardized daily activities | at day the 1st , 4th day of a 4 weeks rehabilitation program.
  Pain intensity evaluation with a 100 mm Visual Analogue Scale (VAS) from 0 to
Percentage of improved patients | at day the 1st , 4th and 5th day of a 4 weeks rehabilitation program.
  Percentage of patients reporting pain improvement of at least 20 mm on the Visual Analogue Scale with the ATLAS device during the 5 standardized daily activities compared to the pain reported without wearing the ATLAS device during the same 5 standardized daily activities (the most intense pain reported during the 5 activities is recorded).
Percentage of patients relieved with the ATLAS device | at day the 1st , 4th and 5th day of a 4 weeks rehabilitation program.
  Percentage of patients wearing the ATLAS device reporting pain intensity less than 30 mm on a 100mm Visual Analogue scale during the 5 standardized daily activities (the most intense pain reported during the 5 activities is recorded).

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Tiffreau, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Swynghedau, CHU, Lille, France